CLINICAL TRIAL: NCT06464302
Title: Investigation of the Effect of Age and Injury Severity on Short-term Intra-hospital Outcomes After Surgical Stabilized Rib Fractures
Status: Recruiting | Type: Observational
Sponsor: University Hospital Muenster (Other)
Responsible Party: Sponsor
Other Study IDs: UKM_UCH_2024_002
Record Dates: First submitted 2024-05-31; First posted 2024-06-18 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2025-06

CONDITIONS: Rib Fractures; Rib Trauma; Rib Fracture Multiple; Thorax; Fracture
Keywords: Surgical stabilisation of rib fractures (SSRF)
MeSH Terms: conditions — Rib Fractures; Fractures, Bone

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Operative: Patients receiving surgical stabilisation of rib fractures (SSRF) by any operative technique
  Interventions: Procedure: Surgical stabilisation of rib fractures (SSRF); Other: Non-operative management of rib fractures
- Non-operative: Patients not receiving surgical stabilisation of rib fractures (SSRF)
  Interventions: Other: Non-operative management of rib fractures

INTERVENTIONS:
Procedure: Surgical stabilisation of rib fractures (SSRF) — Surgical stabilisation of rib fractures using any fixation technique (including but not limited to plate fixation, intramedullary fixation, wire fixation) via any operative approach (including but not limited to open external approach, minimally invasive approach, thoracoscopic approach, thoracotomy approach).
  Groups: Operative
Other: Non-operative management of rib fractures — Any supportive or specific treatment of rib fractures excluding surgical stabilisation of rib fractures. This includes, but is not limited to analgesia, physiotherapy, non-invasive ventilation, mechanical ventilation, oxygen-supplementation

SUMMARY:
The study aims to investigate the effect of surgical stabilisation of rib fractures (SSRF) on clinical outcomes measured during the hospital stay (mortality, days on a mechanical ventilator, intensive care unit and hospital length of stay, rate of complications). Furthermore, the effect of the patients age and overall injury severity on the outcomes after SSRF will be investigated. We hypothesise that the combination of high age and high injury severity will lead to worse outcomes after SSRF.

ELIGIBILITY:
Inclusion Criteria:

* Patients of the University Hospital Muenster
* Coded serial rib fractures (ICD S22.4 and S22.5)
* Treatment for the rib fractures between 2019 and 2023

Exclusion Criteria:

* pathological rib fractures (due to suspected malignancy)

Ages: 0 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The Patients will be sampled from all patients treated in the department for trauma, hand and reconstructive surgery of the university hospital Muenster
Sampling Method: Probability Sample
Enrollment: 700 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
In hospital-mortality | From injury up to initial hospital discharge or death, whichever came first, assessed up to 2 month.
  Mortality rate from injury to initial hospital discharge, binary
Intensive care unit length of stay | From injury up to initial hospital discharge or death, whichever came first, assessed up to 2 month.
  The duration in days a patient spent in the intensive care unit from the time of hospital admission to the time of initial hospital discharge.

SECONDARY OUTCOMES:
Intubation rate | From injury up to initial hospital discharge or death, whichever came first, assessed up to 2 month.
  Proportion of patients intubated at any time
Multi-organ failure | From injury up to initial hospital discharge or death, whichever came first, assessed up to 2 month.
  Rate of Multi-organ failure
Single organ failure | From injury up to initial hospital discharge or death, whichever came first, assessed up to 2 month.
  Rate of single organ failure
Sepsis | From injury up to initial hospital discharge or death, whichever came first, assessed up to 2 month.
  Rate of Sepsis
Lung-failure | From injury up to initial hospital discharge or death, whichever came first, assessed up to 2 month.
  Rate of Lung-failure
Clinical outcome | At the time point of initial hospital discharge or at death, whichever came first, assessed up to 2 month.
  Clinical outcome according to the Glasgow outcome scale (GOS)
Duration of hospital stay | From injury up to initial hospital discharge or death, whichever came first, assessed up to 2 month.
  Duration of hospital stay in days from injury to initial discharge

CONTACTS AND LOCATIONS:
Overall Officials: Steffen Rosslenbroich, PD Dr. med., Study Director — Department for trauma, hand and reconstructive surgery, University hospital Muenster
Locations (1):
- Department for trauma, hand and reconstructive surgery, University hospital Muenster, Münster, North Rhine-Westphalia, Germany

IPD SHARING:
Plan to Share IPD: Undecided